CLINICAL TRIAL: NCT03790683
Title: Intraoperative Warming During Major Surgical Procedures Using the Esophageal Temperature Management System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor funding limitations
Sponsor: Advanced Cooling Therapy, Inc., d/b/a Attune Medical (Industry)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Advanced Cooling Therapy LLC, d/b/a Attune Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TJ Intraoperative warming
Record Dates: First submitted 2018-12-27; First posted 2019-01-02 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Hypothermia Following Anesthesia; Hypothermia; Surgery
Keywords: intraoperative hypothermia; inadvertent hypothermia; perioperative hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: prospective, randomized interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EnsoETM (Experimental): Participants receive esophageal warming. Original study design anticipated esophageal warming in addition to standard of care surface warming from the time they enter the OR until released to the PACU. After 7 patients, protocol was adjusted to specify only esophageal warming unless addition of surface warming was warranted.
  Interventions: Device: EnsoETM; Device: Surface Warming
- Standard of Care (Active Comparator): Participants receive standard of care surface warming from the time they enter the OR until released to the PACU.
  Interventions: Device: Surface Warming

INTERVENTIONS:
Device: EnsoETM — Patients having major surgery will have the EnsoETM device placed after induction of general anesthesia. Addition of standard of care surface warming was specified as optional after first 7 patients.
  Other Names: ECD02, Esophageal Cooling Device
  Arms: EnsoETM
Device: Surface Warming — Forced air warming device will be placed on the patient according to standard practice.
  Other Names: Bair Hugger, forced air blanket

SUMMARY:
The aim of this study is to assess the effectiveness of EnsoETM as a supplemental warming device compared to the standard of care warming practice in patients having major surgery.

DETAILED DESCRIPTION:
Maintaining patient's body temperature is of major importance in patients undergoing surgical procedures and existing methods to warm patients to maintain perioperative normothermia have limitations. This results in as many as half of patients undergoing surgery developing inadvertent hypothermia during and/or after their procedure. The EnsoETM is an Esophageal Temperature Management (ETM) device consisting of a multi-chambered silicone tube connected to a heat exchanger and placed in the esophagus, providing highly efficient heat transfer to a patient. The EnsoETM potentially improves the ability to control patient temperature by eliminating the disadvantages of existing methods while maintaining the functionality of the orogastric tube that it replaces.

The primary objective of this study is to measure the number of degree-hours spent below 37°C intraoperatively and until recovery in the PACU. This measure will be compared between patients having standard management of body temperature to patients having the EnsoETM placed as an additional warming device.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Male or female, ages 18 years and older
* Scheduled for major surgical procedures requiring general anesthesia and with no known contraindication to having an orogastric tube placed for the duration of the surgery
* The time in the OR is expected to last at least 180 minutes

Exclusion Criteria:

* Esophageal strictures (risk of perforation)
* Patients with known esophageal deformity or evidence of esophageal trauma (for example history of esophagectomy, previous swallowing disorders, achalasia, etc.)
* Known ingestion of acidic or caustic poisons within the prior 24 hours.
* Patients with <40 kg of body mass
* Coagulopathy
* Severe facial trauma
* Surgical procedures lasting less than 3 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleen Vernick, DO, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EnsoETM: Participants receive esophageal warming only from the time they enter the OR until released to the PACU.
  EnsoETM: Patients having major surgery will have the EnsoETM device placed after induction of general anesthesia.
Period: Overall Study
Arm/Group | EnsoETM | Standard of Care
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EnsoETM | Standard of Care | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (14.3) | 65.4 (7.4) | 61.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Inadvertent Hypothermia Prevention
Description: Number of degree-hours spent below 37 °C intraoperatively until recovery in the PACU and return to 37°C body temperature.
Time Frame: Time from intubation until extubation, approximately 3-12 hours
Measure: Mean (Standard Deviation); unit: degrees Celsius*hours
Arm/Group | EnsoETM | Standard of Care
Number analyzed (Participants) | 14 | 14
degrees Celsius*hours | 5.85 (.36) | 4.25 (.41)

2. Secondary Outcome: Time From Intubation Until Extubation
Description: Time from intubation until extubation
Time Frame: perioperative, approximately 3-12 hours
Population: Data were not collected and the outcome cannot be reported.
Arm/Group | EnsoETM | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During and up to 24 hours after surgery, a total of approximately 36 hours.
Arm/Group | EnsoETM | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03790683/Prot_SAP_000.pdf